CLINICAL TRIAL: NCT02146144
Title: Prospective, Randomized, Controlled and Single-blind Study Assessing the Benefit/Risk Ratio of Internal Limiting Membrane (ILM) Peeling During Epimacular Membrane (EMM) Surgery
Brief Title: Prospective, Single-blind Study Assessing the Benefit/Risk Ratio of Internal Limiting Membrane (ILM) Peeling During Epimacular Membrane (EMM) Surgery (Peeling)
Acronym: Peeling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC14_0026
Record Dates: First submitted 2014-04-07; First posted 2014-05-23 (Estimated); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Idiopathic Epimacular Membrane
Keywords: Idiopathic epimacular membrane; internal limiting membrane peeling; microscotomas

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- no peeling (No Intervention): where the ILM peeling will not be made
- active peeling (Active Comparator): where the ILM peeling will be made
  Interventions: Procedure: ILM Peeling

INTERVENTIONS:
Procedure: ILM Peeling — common surgical procedure:
  For phakic eyes with cataract • phacoemulsification and implantation of a posterior chamber intraocular lens
  For all patients:
  * Central and peripheral 25 Gauge vitrectomy
  * dissection of the epimacular membrane
  * injection of Membraneblue-Dual® according to protocol, wait of 1 minute with the infusion line closed, and then suction of surplus and washing of the vitreous cavity
  * Intraoperative picture to see the possible spontaneous ILM peeling
  * If no spontaneous ILM peeling, the patient will be randomized at the operating block
  Specific surgical procedure:
  • • Randomization into two groups:
  * Arm 1: "no peeling", where the ILM peeling will not be made
  * Arm 2: "active peeling", where the ILM peeling will be made
  Arms: active peeling

SUMMARY:
The epimacular membrane (EMM) is a degenerative condition associated with age, with a variable impact on vision. Treatment is surgery based and consists of a vitrectomy followed by a peeling of the epimacular membrane using a microgripper. Peeling of the internal limiting membrane (ILM) is an adjuvant action that is now frequently practiced and which is expected to increase the success rate of EMM surgery by reducing the risk of recurrence of EMM. Although ILM peeling does not seem to have an adverse effect on visual acuity, it is not totally without consequence, it involves the risk of histological disorganization of the retina at the origin of one or several microscotomas, which are themselves responsible for a final visual discomfort. These microscotomas, resulting in the perception of somewhat black spots visible near the fixed point or the fixed image, may be highlighted by microperimetry and would be a loss of functional opportunity for the patient.

In addition, recurrence of EMM, which the ILM peeling is supposed to diminish, does not alter the vision in half the patients. Furthermore, for those patients who are functionally affected by any such recurrence, a second epimacular membrane peeling surgery can be done.

The main objective of this study is to compare the difference in microscotoma(s) before surgery and 6 months later, between an "active ILM peeling" group and a "no ILM peeling" group. Given the more invasive nature of ILM peeling, the investigators believe that the rate of microscotomas in these patients is higher than those without peeling.

DETAILED DESCRIPTION:
The visits for this trial are those planned for patients receiving EMM surgical operation, namely:

Selection/Inclusion visit : D-90 to D-7 This visit can be split in two according to the requirements of the investigator and/or the patient.

* Full information about the trial
* Verification of the inclusion and non-inclusion criteria
* Obtaining the signed informed consent (the same day or after a period of reflection)
* Medical and surgical history - *Examination: Visual acuity measured on the ETDRS scale, near vision (Parinaud), spectral domain optical coherence tomography (SD-OCT), microperimetry and pre-operative: "Patient discomfort" questionnaire (Appendix 7), an assessment of the appearance of the lens at the slit lamp, examination of the fundus after pupillary dilation, biomicroscopic examination of the anterior segment, retinal photography.

Surgery visit D0:

* List of all the surgical procedures
* Randomization for ILM peeling or not, in the operating room after dyeing of the ILM by the Membraneblue-Dual® (Picture of the macula). An anonymous video of the surgery will be sent to Nantes for centralized processing of the analysis of the EMM's grip areas.

To avoid bias, the follow-up visits will be made by an ophthalmologist and/or an orthoptist who will not know what action has been performed.

Follow-up visit M1 (1 month after the surgery ± 7 days)

* Examination: Visual acuity measured on the ETDRS scale, near vision (Parinaud), spectral domain optical coherence tomography (SD-OCT), Microscopic examination of the eye, microperimetry, fundus photography and post-operative "Patient discomfort" questionnaire (Appendix 8). Biomicroscopic examination of the anterior segment, retinal photography.
* AE

Follow-up visit M6 (6 months after the surgery ± 15 days)

* Examination: Visual acuity measured on the ETDRS scale, near vision (Parinaud), spectral domain optical coherence tomography (SD-OCT), Microscopic examination of the eye, microperimetry, fundus photography and post-operative: "Patient discomfort" questionnaire (Appendix 8). Biomicroscopic examination of the anterior segment, retinal photography.
* AE End of study visit M12 (12 months after the surgery ± 15 days)
* Examination: Visual acuity measured on the ETDRS scale, near vision (Parinaud), spectral domain optical coherence tomography (SD-OCT), Microscopic examination of the eye, microperimetry, fundus photography and post-operative "Patient discomfort" questionnaire (Appendix 8), Biomicroscopic examination of the anterior segment, retinal photography.
* AE

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years old) and female without childbearing potential or active contraception (intra-uterine device, contraceptive pill or contraceptive implant).
* Patients with an idiopathic symptomatic epimacular membrane; for patients with both eyes affected, the eye treated in the protocol will be the one which is most severely affected.
* Pseudophakic patients with transparent posterior capsule or open capsule or lensed patients with age-related cataracts
* Patients with social security
* Patients able to understand and follow the trial instructions
* Patients who have signed an informed consent

Exclusion Criteria:

* Patient with other retinal pathologies such as age related macular degeneration ("AMD"), retinal vein occlusion, diabetic retinopathy, glaucoma with macular visual field defect
* Patients with uveitis or history of uveitis
* Patients with any recent eye injuries or eye surgeries (<6 months)
* Patients participating in interventional clinical trial
* Pregnant or breast feeding women
* Vulnerable people : persons deprived of liberty; under trusteeship or under curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2014-09-09 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2022-03-14 (Actual)

PRIMARY OUTCOMES:
the difference in microscotomas between the inclusion visit and the visit at 6 months after surgery. | 6 months
  Analysis of the primary endpoint: the main criterion is the difference between the number of microscotomas measured before surgery and the number of microscotomas measured at 6 months (number between 0 and 29).
  The mean difference will be calculated in each of two groups and compared using a mixed model of linear regression to take into account the stratification of the randomization at the center (the center will be considered as a random effect)

SECONDARY OUTCOMES:
Study of anatomical and functional changes of the retina | 12 months
  Number and types of microscotomas by microperimetry (before and after surgery)
Study the rate of EMM recurrence (at M12) between the 2 groups. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ramin Tadayoni, Pr, Principal Investigator — Hôpital Lariboisière, AP-HP; Catherine Creuzot-Garchet, Pr, Principal Investigator — Centre Hospitalier Universitaire Dijon; Yannick Le Mer, Pr, Principal Investigator — Fondation Ophtalmologique A. de Rothschild
Locations (6):
- France (6):
  - CHU de Dijon, Dijon
  - Clinique Sourdille, Nantes
  - CHU de Nantes, Nantes
  - Fondation Ophtalmologique A. de Rothschild, Paris
  - Hôpital Lariboisière (AP-HP), Paris
  - Polyclinique de l'atlantique, Saint-Herblain

REFERENCES:
- [Derived] Ducloyer JB, Eude Y, Volteau C, Lebreton O, Bonissent A, Fossum P, Tadayoni R, Creuzot-Garcher CP, Le Mer Y, Perol J, Fortin J, Jobert A, Billaud F, Ivan C, Poinas A, Weber M; CFSR Research Net. Pros and cons of internal limiting membrane peeling during epiretinal membrane surgery: a randomised clinical trial with microperimetry (PEELING). Br J Ophthalmol. 2024 Dec 17;109(1):119-125. doi: 10.1136/bjo-2023-324990. PMID 38901960
- [Derived] Ducloyer JB, Ivan J, Poinas A, Lebreton O, Bonissent A, Fossum P, Volteau C, Tadayoni R, Creuzot-Garchet C, Le Mer Y, Perol J, Fortin J, Chiffoleau A, Billaud F, Ivan C, Weber M. Does internal limiting membrane peeling during epiretinal membrane surgery induce microscotomas on microperimetry? Study protocol for PEELING, a randomized controlled clinical trial. Trials. 2020 Jun 8;21(1):500. doi: 10.1186/s13063-020-04433-9. PMID 32513229